CLINICAL TRIAL: NCT03629756
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of Immunotherapy Combinations in Participants With Advanced Malignancies
Brief Title: A Study to Evaluate the Safety and Tolerability of Immunotherapy Combinations in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-5 (AB928CSP0005)
Record Dates: First submitted 2018-07-17; First posted 2018-08-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Breast Cancer; Colorectal Cancer; Melanoma; Bladder Cancer; Ovarian Cancer; Endometrial Cancer; Merkel Cell Carcinoma; GastroEsophageal Cancer; Renal Cell Carcinoma; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Colorectal Neoplasms; Melanoma; Urinary Bladder Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Merkel Cell; Carcinoma, Renal Cell | interventions — zimberelimab

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): 3+3 design, including a DLT evaluation period. Etrumadenant RP2D will be determined in this part with escalating doses of oral etrumadenant in combination with a fixed dose of IV zimberelimab.
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab
- Dose Expansion-advanced clear-cell RCC (Experimental): Etrumadenant at RP2D + zimberelimab
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab
- Dose Expansion-mCRPC (Experimental): Etrumadenant at RP2D + zimberelimab
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab

INTERVENTIONS:
Drug: Etrumadenant — Etrumadenant is an A2aR and A2bR antagonist.
  Other Names: AB928
Drug: Zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody.
  Other Names: AB122

SUMMARY:
This is a Phase 1, open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) and clinical activity of etrumadenant (AB928) in combination with zimberelimab (AB122) (an anti-PD-1 antibody) in participants with advanced malignancies.

DETAILED DESCRIPTION:
In the dose-escalation phase, escalating doses of etrumadenant in combination with zimberelimab will be assessed in participants with advanced malignancies. Eligible participants will receive oral administration of etrumadenant as well as IV infusion of zimberelimab. The recommended Phase 2 dose (RP2D) of etrumadenant will be determined upon completion of the dose-escalation phase.

In the dose-expansion phase, etrumadenant at RP2D in combination with zimberelimab may be assessed in participants with advanced clear-cell renal cell carcinoma (RCC) or metastatic castrate-resistant adenocarcinoma of the prostate (mCRPC).

Overall duration of treatment will depend on how well the treatment is tolerated. Treatment may continue until unacceptable toxicity or progressive disease or other reasons specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years
2. Must have at least 1 measurable lesion per RECIST v1.1.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Must have received standard of care, including potentially curative available therapies or interventions.
5. Confirm that an archival tissue sample is available and ≤ 6 months old; if not, a new biopsy of a tumor lesion must be obtained. Biopsy must not put participant at undue risk and the procedure must not be more invasive than a core biopsy.
6. Adequate organ and marrow function

   Dose escalation only:
7. Pathologically confirmed non-small cell lung cancer, squamous cell carcinoma of the head and neck, renal cell carcinoma, breast cancer, colorectal cancer, melanoma, bladder cancer, ovarian cancer, endometrial cancer, Merkel cell carcinoma, or gastroesophageal cancer that is metastatic, advanced or recurrent with progression for which no alternative or curative therapy exists or standard therapy is not considered appropriate by the participant and treating physician (reason must be documented in medical records).

   Dose expansion only:
8. Participants with advanced clear-cell RCC or mCRPC.9. Clear-cell RCC participants may have received up to 2 prior lines of therapy, one of which must have included an anti-PD-(L)1 based therapy and must not have progressed within 16 weeks during an anti-PD-(L)1 therapy.
9. mCRPC participants must have progressed during or following treatment with an androgen synthesis inhibitor, and have also had one prior line of a taxane-containing regimen or the physician and participant consider the taxane-containing regimen to be inappropriate.
10. mCRPC participants must be naive to any immunotherapy (including but not limited to anti-PD-(L)1 or anti-CTLA-4 antagonists, sipuleucel-T, etc.).

Exclusion Criteria:

1. Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of investigational product.
2. Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of investigational product hazardous (eg, interstitial lung disease, active infections requiring antibiotics, recent hospitalization with unresolved symptoms) or obscure the interpretation of toxicity determination or AEs, or concurrent medical condition requiring the use of immunosuppressive medications or immunosuppressive doses of systemic or absorbable topical corticosteroids.
3. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
4. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 90 days after the last dose of etrumadenant in combination with zimberelimab.
5. Any active or documented history of autoimmune disease, or history of a syndrome that required systemic steroids or immunosuppressive medications, except for vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study.
6. Prior malignancy active within the previous year except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, breast, or prostate cancer.
7. Dose escalation: Prior treatment with an anti-PD-L1, anti-PD-1, anti-CTLA-4, or other immune checkpoint inhibitor or agonist as a monotherapy or in combination;
8. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before investigational product administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events | From first dose date to 90 days after the last dose (approximately 3 years)
  Safety will be assessed by monitoring adverse events and clinically relevant changes in Eastern Cooperative Oncology Group (ECOG) performance status, 12 lead Electrocardiogram (ECG), vital signs, physical examination and clinical laboratory results.
Percentage of participants who experience a Dose Limiting Toxicity | From first study treatment administration through Day 28

SECONDARY OUTCOMES:
Etrumadenant Peak Serum Concentration: Cmax | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 and 90 days post last dose (approximately 7 months)
Zimberelimab Peak Serum Concentration: Cmax | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 and 90 days post last dose (approximately 7 months)
Etrumadenant Time of Peak Concentration: Tmax | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 and 90 days post last dose (approximately 7 months)
Zimberelimab Time of Peak Concentration: Tmax | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 and 90 days post last dose (approximately 7 months)
Percentage of participants with anti-drug antibodies to zimberelimab | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months), at end of treatment, and 30 and 90 days post last dose (approximately 7 months)
Progression Free Survival (PFS) | From start of treatment up to the first occurrence of progressive disease or death from any cause (approximately 1-3 years)
  PFS as determined by Investigator according to Prostate Cancer Working Group 3 (PCWG3) for prostate adenocarcinoma and per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for all other tumor types
Overall Survival (OS) | From study start of treatment up to death from any cause (approximately 1-3 years)
  OS as determined by the Investigator according to PCWG3 for prostate adenocarcinoma and per RECIST v1.1 for all other tumor types
Duration of Response (DOR) | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (approximately 1-3 years)
  DOR as determined by the Investigator according to PCWG3 for prostate adenocarcinoma and per RECIST v1.1 for all other tumor types
Percentage of Participants with Disease Control | From study enrolment until disease progression or loss of clinical benefit (approximately 1-3 years)
  Disease Control (complete response, partial response, or stable disease) for >6 months as determined by the Investigator per PCWG3 for prostate adenocarcinoma and per RECIST v1.1 for all other tumor types
Percentage of participants with Objective Response | From study enrolment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 1-3 years)
  Objective Response as determined by Investigator according to PCWG3 for prostate adenocarcinoma and per RECIST v1.1 for all other tumor types

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (15):
- United States (12):
  - Scottsdale Healthcare Hospitals dba HonorHealth, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Rocky Mountain Cancer Centers (Midtown), Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - QUEST Research Institute, Royal Oak, Michigan
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Texas Oncology, P.A. - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, P.A. - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Medical Oncology Associates dba Summit Cancer Centers, Spokane, Washington
- Australia (3):
  - St. George Private Hospital, Kogarah, New South Wales
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Cabrini Health Limited, Malvern

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-5 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=ARC-5